CLINICAL TRIAL: NCT05192603
Title: Comparison in the Effects and Mechanisms Between Low Fermentable-, Oligo-, di-, and Monosaccharides and Polyols (FODMAP) and Starch- and Sucrose-reduced Diet (SSRD) in Irritable Bowel Syndrome (IBS)
Brief Title: Comparison Between Low FODMAP and SSRD in IBS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Bodil Ohlsson, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-2021
Record Dates: First submitted 2021-11-29; First posted 2022-01-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS; low FODMAP; SSRD
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, open study for dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention with Low FODMAP (Experimental): The participants are given oral and written instructions on which diet that contains low contents of FODMAP.
  Interventions: Dietary Supplement: low FODMAP or SSRD
- Dietary intervention with SSRD (Experimental): The participants are given oral and written instructions on which diet that contains SSRD.
  Interventions: Dietary Supplement: low FODMAP or SSRD

INTERVENTIONS:
Dietary Supplement: low FODMAP or SSRD — The participants are given oral and written information about each diet. No food is delivered from the investigator to the participant

SUMMARY:
The aim of the present study is to compare the efficiency of low FODMAP and SSRD to reduce symptoms in IBS, and to study the mechanisms and consequences of the two diets.

DETAILED DESCRIPTION:
The investigator will perform a study on 200 subjects with verified irritable bowel syndrome (IBS). Participants will be recruited from the clinic of Gastroenterology or Internal medicine as well as primary health care centers. At the start of the study, participants will complete protocols concerning Rom IV criteria (to validate that the IBS criteria are ful-filled) as well as IBS symptom rating scales irritable bowel syndrome-symptoms severity scores (IBS-SSS) and visual analog scale for irritable bowel syndrome (VAS-IBS). The Item Health Survey 1.0 (distributed by RAND), RAND-36, includes the same items as those in the Short-Form Health Survey (SF-36), and evaluates the quality of Life. SCOFF is a brief questionnaire that asks the five questions about eating disturbances (Do you make yourself Sick because you feel uncomfortably full? Do you worry you have lost Control over how much you eat? Have you recently lost more than One stone in a 3 month period? Do you believe yourself to be Fat when others say you are too thin? Would you say that Food dominates your life?). Participants will be examined by an investigator who will complete protocols of clinical data. Blood and fecal samples will be collected by the investigator.

Study participants will thereafter be randomized to receive either low FODMAP (Fermentable, Oligo-, Di-, Mono-saccharides And Polyols) diet (n=100), or a SSRD diet (starch ans sucrose-reduced diet) (n=100). After 4 weeks of dietary intervention, there will be a follow-up where blood and fecal samples are once again collected. At this point in time, participants will also fill in IBS symptom rating scales again.

The participants are then free to eat whatever they want to, and another 5 months later, they will be examined again, the same protocols will be completed, and blood and fecal samples are collected.

The investigator will use samples from baseline, 4 weeks and 6 months, for genetic/epigenetic (including genomic-wide association studies), metabolomics, proteomics, nutritional data, gut microbiota, and inflammatory parameter analyses.

Statistics

The investigator will use Mann-Whitney U-test and Wilcoxon test to study differences in the above-mentioned parameters between the two treatment groups, as well as before and after dietary intervention, respectively. For analyses of genetic/epigenetics, metabolomics, proteomics, and microbiota, the investigator will use bioinformatics and biostatistics.

ELIGIBILITY:
Inclusion Criteria:

* Verified IBS according to Rom IV criteria.

Exclusion Criteria:

* Serious mental disease
* Serious somatic disease
* Abuse
* Inability to understand the Swedish language
* Already on a diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency on bowel and extra-intestinal symptoms | 4 weeks dietary intervention
  To assess bowel symptoms and extra-intestinal symptoms after the dietary interventions by evaluation of irritable bowel syndrome-symptom severity score (IBS-SSS). This questionnaire contains VAS scales ranging from 0-100 where a higher score means worse symptoms.
Efficiency on bowel and extra-intestinal symptoms | A follow-up 5 months after the end of the intervention
  To assess bowel symptoms and extra-intestinal symptoms after the dietary interventions by evaluation of IBS-SSS. This questionnaire contains VAS scales ranging from 0-100 where a higher score means worse symptoms.
Efficiency on bowel symptoms | 4 weeks dietary intervention
  To assess bowel symptoms after the dietary interventions by evaluation of visual analog scale for irritable bowel syndrome (VAS-IBS). This questionnaire contains VAS scales ranging from 0-100 where a higher score means worse symptoms.
Efficiency on bowel symptoms | A follow-up 5 months after the end of the intervention
  To assess bowel symptoms after the dietary interventions by evaluation of visual analog scale for irritable bowel syndrome (VAS-IBS). This questionnaire contains VAS scales ranging from 0-100 where a higher score means worse symptoms.

SECONDARY OUTCOMES:
Effects on plasminogen activator inhibitor-1 (PAI-1) | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze plasminogen activator inhibitor-1 (PAI-1) by enzyme-linked immunosorbent assay (ELISA) to see and compare the effects of the two different diets.
Effects on C-peptide | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze C-peptide by enzyme-linked immunosorbent assay (ELISA) to see and compare the effects of the two different diets.
Effects on insulin | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze insulin by enzyme-linked immunosorbent assay (ELISA) to see and compare the effects of the two different diets.
Effects on leptin | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze leptin by enzyme-linked immunosorbent assay (ELISA) to see and compare the effects of the two different diets.
Effects on gastric inhibitory peptide (GIP) | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze GIP by enzyme-linked immunosorbent assay (ELISA) to see and compare the effects of the two different diets.
Effects on visfatin | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze visfatin by mesoscale to see and compare the effects of the two different diets.
Effects on ghrelin | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze ghrelin by mesoscale to see and compare the effects of the two different diets.
Effects on gut microbiota by whole genome sequencing of feces | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze fecal microbiota by whole genome sequencing to see and compare the effects of the two different diets
Effects on microRNA | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze microRNA to see and compare the effects of the two different diets
Effects on DNA methylation | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze DNA methylation to see and compare the effects of the two different diets
Effects depending on genetics | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze sucrase-isomaltase (SI) genes to see if the genetic profile hais of importance for the clinical effect of the two diets
Effects on vitamin A | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of vitamin A in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on vitamin B | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of vitamin B in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on vitamin C | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of vitamin C in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on vitamin D | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of vitamin D in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on phosphorous | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of phosphorous in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on zinc | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of zinc in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on magnesium | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of magnesium in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on albumin | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze values of albumin in blood before and after the study to compare the effects on the nutritional status by the two diets.
Effects on metabolomics and proteomics | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze metabolomics and proteomics in blood to see and compare the effects of the two different diets
Effects on quality of life by RAND-36 (comprehensive short-form generic profile for health-related quality of life (HRQoL)) | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze how the two different diets influence quality of life, measured by RAND-36, to compare the effects of the two different diets. RAND-36 is comprised of 36 items on 5-point Likert scale, the higher score the better quality of life, that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
Effects on eating disturbances | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze how the two different diets influence eating disturbances measured by SCOFF, to compare the effects of the two different diets. SCOFF contains 5 questions answered by "yes" or "no": 1) Do you make yourself Sick because you feel uncomfortably full?, 2) Do you worry that you have lost Control over how much you eat?, 3)Have you recently lost more than One stone (14 lb) in a 3-month period?, 4)Do you believe yourself to be Fat when others say you are too thin?, and 5) Would you say that Food dominates your life?
Effects on healthcare consumption | 4 weeks dietary intervention, with a follow-up after another 5 months
  The investigator will analyze how the two different diets influence healthcare consumption by asking the participants about how many times they have visited a Healthcare giver before, during and after the study, to compare the effects of the two different diets

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Ohlsson, Professor, Principal Investigator — Department of Internal Medicine; Bodil Roth, PhD, Study Chair — Department of Internal Medicine
Locations (1):
- Deartment of INternal Medicine, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth B, Ohlsson B. Overweight and vitamin D deficiency are common in patients with irritable bowel syndrome - a cross-sectional study. BMC Gastroenterol. 2024 Sep 3;24(1):296. doi: 10.1186/s12876-024-03373-x. PMID 39227769
- [Derived] Roth B, Ohlsson B. Challenges of recruitment processes to a randomized dietary trial in irritable bowel syndrome. F1000Res. 2024 Jun 24;13:323. doi: 10.12688/f1000research.147710.2. eCollection 2024. PMID 38939366
- [Derived] Roth B, Ohlsson B. A starch- and sucrose-reduced diet may lead to improvement of intestinal and extraintestinal symptoms in more conditions than irritable bowel syndrome and congenital sucrase-isomaltase deficiency. Nutrition. 2024 Jan;117:112254. doi: 10.1016/j.nut.2023.112254. Epub 2023 Oct 8. PMID 37924624